CLINICAL TRIAL: NCT06846307
Title: The Effect of Mannitol Volume Administration with Changes in Osmolarity in Traumatic Brain Injury: an Observational Study
Brief Title: The Effect of Mannitol Volume with Changes in Osmolarity in Traumatic Brain Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Taufik Saputra, Resident of Anesthesiology and Intensive Care, Medical Doctor, Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1554/EC/KEPK-RSDK/2023
Record Dates: First submitted 2025-02-04; First posted 2025-02-26 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia; Traumatic Brain Injury
Keywords: brain injury; intracranial pressure; mannitol; neurocritical care; osmolarity; trauma
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Wounds and Injuries | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mannitol 1 (Active Comparator): mannitol 3x125 cc
  Interventions: Drug: Mannitol
- Mannitol 2 (Active Comparator): Mannitol 2x250 cc
  Interventions: Drug: Mannitol
- Mannitol 3 (Active Comparator): Mannitol 3x250 cc
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Mannitol — mannitol administration across all three dosages (3x125 cc, 2x250 cc, 3x250 cc) given as an IV drip for 15-20 minutes
  Other Names: Otsu-Mannitol 20

SUMMARY:
This observational study is designed to research the effect of mannitol volume administration with changes in osmolarity in patients with traumatic brain injury to guide the safe use of mannitol in these patients.

DETAILED DESCRIPTION:
This study used an analytic observational design with a prospective cohort approach to evaluate the relationship between mannitol administration volume and changes in osmolarity in TBI patients at Dr. Kariadi Central General Hospital, Semarang, Indonesia. The study included 32 non-operative TBI patients admitted to the Emergency Department (ED) and inpatient wards from November 2023 to January 2024. Samples were selected using a consecutive sampling method based on the inclusion criteria. The independent variable in this study was the volume of mannitol administered (3x125 cc, 2x250 cc, 3x250 cc; each 250 cc contains 50g mannitol) given as an IV drip for 15-20 minutes, while the dependent variable was blood osmolarity (mOsm/L).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-40 years
* Glasgow Coma Scale (GCS) score indicating mild (14-13) or moderate (12-10)

Exclusion Criteria:

* Renal impairment
* Multiple trauma with bleeding shock
* Diabetes mellitus

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Osmolarity | At baseline (before administration) and subsequently at 6 hours and 24 hours post-administration
  Blood osmolarity (mOsm/L)

CONTACTS AND LOCATIONS:
Overall Officials: Aria P Hayanto, Sp.An-TI, Study Director — Universitas Diponegoro
Locations (1):
- Dr. Kariadi Central General Hospital, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No